CLINICAL TRIAL: NCT00000598
Title: Diet and Exercise for Elevated Risk (DEER)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Purpose: Prevention
Other Study IDs: 501; R01HL045733 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia | interventions — Diet, Fat-Restricted; Exercise

INTERVENTIONS:
Behavioral: diet, fat-restricted
Behavioral: exercise

SUMMARY:
To determine the effect in men and postmenopausal women with elevated LDL-cholesterol and low HDL-cholesterol of an exercise regimen with or without the National Cholesterol Education Program (NCEP) Step Two diet compared to usual care control group on HDL- and LDL-cholesterol.

DETAILED DESCRIPTION:
BACKGROUND:

The NCEP is a major public education program providing advice to physicians and the public on management and prevention of coronary heart disease. However, data supporting the advice are derived primarily from middle-aged men, with less data available for women and older individuals. Furthermore, there have been recent reports that when low saturated fat diets such as the NCEP Step One and NCEP Step Two diets, are followed, HDL-cholesterol is lowered as well as LDL-cholesterol.

DESIGN NARRATIVE:

Randomized, controlled, factorial design powered for men and women separately. One hundred eighty postmenopausal women, 45 through 64 years of age, and 197 men, 30 through 64 years of age, who had low high-density lipoprotein (HDL) cholesterol levels (< or =59 mg per deciliter in women and < or =44 mg per deciliter in men) and moderately elevated levels of low-density lipoprotein (LDL) cholesterol (>125 mg per deciliter but <210 mg per deciliter in women and >125 mg per deciliter but <190 mg per deciliter in men) were enrolled. The subjects were randomly assigned to aerobic exercise, the NCEP Step 2 diet, or diet plus exercise, or to a control group, which received no intervention. The four interventions were delivered for one year: usual care (written dietary materials only with delayed intervention optional), exercise only (supervised, progressive aerobic exercise program at least three times per week), diet only (group and individual dietary instruction on the NCEP Step One/Step Two diet delivered by registered dietitians), and diet plus exercise. At baseline and at the end of one year, measurements were made of blood lipids and lipoproteins, plasma glucose and insulin, glucose tolerance, blood pressure, body composition through hydrostatic weighing and waist and hip circumterences, aerobic fitness (VO2 max), and five unannounced 24-hr. recalls. The primary outcomes measured was HDL-cholesterol, major secondary endpoints included LDL-C, LDL-C/HDL-C ratio, and triglycerides.

ELIGIBILITY:
Men with with LDL-cholesterol of 125-189 mg/dL and HDL-cholesterol below or equal to 44 mg/dL, and postmenopausal women, age 45 to 64, with LDL-cholesterol of 125 to 209 mg/dL and HDL-cholesterol below or equal to 59 mg/dL.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1991-08; Study Completion 1996-08

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wood — Stanford University

REFERENCES:
- [Background] Stefanick ML, Mackey S, Sheehan M, Ellsworth N, Haskell WL, Wood PD. Effects of diet and exercise in men and postmenopausal women with low levels of HDL cholesterol and high levels of LDL cholesterol. N Engl J Med. 1998 Jul 2;339(1):12-20. doi: 10.1056/NEJM199807023390103. PMID 9647874